CLINICAL TRIAL: NCT04818242
Title: Randomized Controlled Trial To Assess the Benefits of Dexcom Continuous Glucose Monitoring With Glucose Telemetry System for the Management of Diabetes in Long-term Care Setting: The CGM-GTS in Long-term Care
Brief Title: Dexcom Continuous Glucose Monitoring in Long-term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001529
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
Keywords: Continuous glucose monitoring; Glucose telemetry system; Long term care
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- POC testing with Blinded CGM (Standard of Care) (Active Comparator): Patients in the standard of care study arm will wear a blinded CGM and receive POC testing before meals and bedtime, with providers adjusting oral agents or insulin dose based on POC results.
  Interventions: Diagnostic Test: POC Blood Glucose Test + Blinded CGM
- Dexcom CGM with Glucose Telemetry System (CGM-GTS) (Experimental): Patients in the intervention CGM study arm will have a single daily fasting POC testing and will wear a real-time Dexcom G6 with GTS, and providers will adjust oral or insulin therapy based on CGM-GTS profile information.
  Interventions: Device: Dexcom G6 CGM with GTS

INTERVENTIONS:
Device: Dexcom G6 CGM with GTS — CGM sensor will be placed after consent. Glucose values obtained from the CGM sensor will be sent to the CGM transmitter by Bluetooth technology and Dexcom Share2 software application to a smart phone that serves as an intermediate-transmitting (routing) device. Glucose values from the smart phone will be transmitted wirelessly to a table computer (I-Pad) using the Dexcom Follow application. Information on the CGM will activate an alarm in case of hypoglycemia or hyperglycemia events. Hypoglycemia alarm will be set to < 85 mg/dl (for prevention for low blood glucose levels). Nursing staff will be instructed to provide 15 grams of carbohydrates in response to a hypoglycemia alarm.The hyperglycemia alarm will be set at 300 mg/dl. If this occurs, the nursing staff will assess clinical status and perform a POC glucose testing to confirm glucose values. If blood glucose (BG) > 300 mg/dl, nursing staff will communicate the high glucose value to the primary care team.
  Other Names: Dexcom Glucose Telemetry System
  Arms: Dexcom CGM with Glucose Telemetry System (CGM-GTS)
Diagnostic Test: POC Blood Glucose Test + Blinded CGM — Point of Care (POC) testing before meals and bedtime (standard of care). For the control group, participants will also get a CGM sensor (blinded CGM). CGM alarms are turned off, however if the POC is found to be between <80 mg/dl by POC, 15 grams of carbohydrates will be given as a preventive measurement for hypoglycemia (standard of care).
  Other Names: Standard of care capillary glucose test and blinded CGM
  Arms: POC testing with Blinded CGM (Standard of Care)

SUMMARY:
The goal of this study is to determine whether the use of Dexcom Continuous Glucose Monitoring with Glucose Telemetry System (CGM-GTS) with hypoglycemia alarm will facilitate diabetes treatment and reduce the risk of hypoglycemia in insulin and non-insulin treated patients with type 2 diabetes (T2D) in long-term care facilities, when compared to standard of care using capillary point of care testing.

DETAILED DESCRIPTION:
The prevalence of diabetes increases with age, and it is estimated that more than 20% of older adults aged 65-75 years and 40% of adults over 80 years of age have diabetes. The prevalence of diabetes in older adults is expected to increase due to longer life expectancy and improvements in care. The estimated prevalence of diabetes in subacute and long-term skilled nursing care facilities is reported to be around 20% to 34% and, in parallel to the increasing geriatric population, the number of long-term care (LTC) admissions is expected to rise.

The goals of diabetes care in older adults and patients in subacute and long-term skilled nursing care facilities include control of hyperglycemia and its symptoms, prevention and treatment of diabetic complications, and maintenance or improvement of general health status. Studies in hospitalized patients with diabetes have shown that improvement in glucose control can reduce complications and are cost savings, however, no prospective studies have determined the impact of improving glucose control on clinical outcome in subacute and long-term skilled nursing care facilities. The management of diabetes in LTC residents is similar to that recommended for ambulatory patients with diabetes, however, several factors complicate the management of hyperglycemia in this population. LTC residents tend to be older and to have higher rates of comorbidities associated with aging such as functional disability, hypertension, coronary artery disease, cerebrovascular events, depression, cognitive impairment, urinary incontinence, and higher risk of falls. In addition, they often experience changes in nutritional intake, which increase the risk of hypoglycemia.

Current guidelines and position statements on diabetes management in older adults are based on consensus opinions or from extrapolations from studies involving middle-aged patients with diabetes. The American Diabetes Association guidelines recommend that older adults who are functional, cognitively intact, and have longer life expectancy should receive diabetes care with goals similar to those developed for younger adults. In these subjects, a HbA1c level <7.5%, a fasting glucose between 90-130 mg/dl, and a random glucose <180 mg/dl is recommended. Less intensive goals are recommended for patients with advanced complications, life-limiting comorbid illness, or cognitive impairment. Other organizations including the American Geriatric Society, European Diabetes Working Party for Older People guidelines, International Association of Gerontology and Geriatrics, the European Diabetes Working Party for Older People recommend a target HbA1c of <7.5% for patients without major comorbidities while a higher target of 7.6-8.5% is proposed for frail patients with high risk of hypoglycemia. These guidelines highlight the importance of improved glucose control and avoidance of side effects and hypoglycemia, as they are associated with increased risk of complications and mortality in patients with diabetes.

Bedside capillary point of care (POC) glucose monitoring is the standard of care to assess glycemic control in the hospital and in LTC facilities. POC testing is usually performed before meals and at bedtime. Continuous glucose monitoring (CGM) measures interstitial glucose every 5-15 minutes, thus providing a more complete glycemic profile during 24-hours than POC testing. This study is a randomized clinical trial to assess the impact of glucose control and hypoglycemia reduction with the use of real time CGM with an alarm system to prevent hypoglycemia and facilitate the care of insulin and non-insulin treated patients with T2D in subacute and long-term skilled nursing care facilities. The results of this study have great potential to impact and facilitate care and to change current clinical guidelines in the management of older adults with diabetes in subacute and LTC facilities.

Residents with T2D in subacute and long-term skilled nursing care facilities treated with insulin and/or insulin-secretagogues will be randomized to a standard of care group with POC testing or to real time Dexcom CGM with GTS until discharge or for up to 60 days of admission (whichever comes sooner). Participants in the standard of care group will wear a blinded CGM and receive POC testing before meals and bedtime, with providers adjusting oral agents or insulin dose based on POC results. Participants in the intervention CGM group will have a single daily fasting POC testing and will wear a real-time Dexcom G6 with GTS, and providers will adjust oral or insulin therapy based on CGM-GTS profile information.

ELIGIBILITY:
Inclusion Criteria:

* Males and females admitted to subacute and long-term skilled nursing care facilities.
* Known history of T2D treated with insulin or insulin secretagogues with or without additional oral antidiabetic agents, short- and long-acting glucagon-like peptide-1 receptor agonists (GLP-1 RA).
* Patients with an expected long-term care facility length-of-stay > 1 week.

Exclusion Criteria:

* Patients expected to require MRI procedures during admission.
* Patients with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), corticosteroid therapy, end-stage renal disease (dialysis), or anasarca (massive peripheral edema).
* Female subjects who are pregnant or breast-feeding at time of enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - A.G. Rhodes, Atlanta, Georgia
  - Emory Wesley Woods Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the results reported in publications from this study (including text, tables, figures, and appendices) will be available for sharing with other researchers who provide a methodologically sound proposal. Individual participant data will be available for sharing for the purpose of achieving the aims in the approved proposal.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing beginning 6 months after publication of the results from this study and ending 5 years after the results from this study were published.
Access Criteria: Proposals should be directed to geumpie@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Wesley Woods Hospital and A.G. Rhodes nursing home in Atlanta, Georgia. Participant enrollment began April 19, 2021 and all follow-up assessments were completed by October 21, 2022.
Groups:
- Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm): Patients in the standard of care study arm wearing a blinded continuous glucose monitoring (CGM) and receiving point-of-care (POC) testing before meals and bedtime, with providers adjusting oral agents or insulin dose based on POC results.
- Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS): Patients in the continuous glucose monitoring (CGM) with glucose telemetry system (CGM-GTS) study arm having a single daily fasting POC testing and wearing a real-time Dexcom G6 with GTS, with providers adjusting oral or insulin therapy based on CGM-GTS profile information.
Period: Overall Study
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Started | 50 | 50
Completed | 50 | 47
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes participants who completed the study.
Groups:
- Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm): Patients in the standard of care study arm wearing a blinded CGM and receiving POC testing before meals and bedtime, with providers adjusting oral agents or insulin dose based on POC results.
- Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS): Patients in the CGM-GTS study arm having a single daily fasting POC testing and wearing a real-time Dexcom G6 with GTS, with providers adjusting oral or insulin therapy based on CGM-GTS profile information.
- Total: Total of all reporting groups
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS) | Total
Number analyzed (Participants) | 50 | 47 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.5 (10.6) | 75.0 (11.8) | 74.7 (11.0)
Age, Customized [Count of Participants; unit: Participants]
  Age 70 or greater | 32 | 31 | 63
  Age less than 70 | 18 | 16 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 14 | 18 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 47 | 97
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (7.3) | 29.9 (8.6) | 29.6 (7.9)
HbA1c [Mean (Standard Deviation); unit: percent of RBCs with glycated hemoglobin] | 8.14 (2.5) | 7.97 (1.9) | 8.06 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Hypoglycemia (BG<70 mg/dL)
Description: The number of participants with hypoglycemia detected, where hypoglycemia is defined as blood glucose (BG) of less than 70 mg/dL.
Time Frame: During hospitalization (up to 60 days of admission)
Population: POC data is unavailable for one participant in the POC study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 49 | 47
Participants | 4 | 9

2. Primary Outcome: Number of Participants Experiencing Clinically Significant Hypoglycemia (BG<54 mg/dL)
Description: Clinically significant hypoglycemia is defined as blood glucose levels less than 54 mg/dL.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
Participants | 0 | 1

3. Primary Outcome: Time in Range (TIR) Between 70-180 mg/dL
Description: Glycemic control is measured by time that blood glucose levels are in the range of 70 to 180 mg/dL.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
percentage of time | 48.8 (28.0) | 53.4 (30.2)

4. Secondary Outcome: Number of Events of Nocturnal Hypoglycemia
Description: The average number of events of nocturnal hypoglycemic events across all participants for BG < 70 mg/dL and <54 mg/dL occurring between 22:00 and 06:00.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
events
  Blood glucose <70 mg/dL | 0.42 (1.23) | 0.55 (1.54)
  Blood glucose <54 mg/dL | 0.28 (0.88) | 0.19 (0.77)

5. Secondary Outcome: Number of Hypoglycemia Events
Description: The total number of events of hypoglycemia events (BG <70 mg/dL and <54 mg/dL) across participants.
Time Frame: During hospitalization (up to 60 days of admission)
Population: POC data is unavailable for one participant in the POC study arm.
Measure: Number; unit: events
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 49 | 47
events
  Blood glucose <70 mg/dL | 4 | 13
  Blood glucose <54 mg/dL | 0 | 1

6. Secondary Outcome: Time in Hypoglycemia (BG<70 mg/dL)
Description: The percent of time in hypoglycemia, defined as blood glucose level <70 mg/dL, is assessed.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
percentage of time | 1.18 (3.5) | 0.83 (2.6)

7. Secondary Outcome: Percent of Time in Hypoglycemia (BG<54 mg/dL)
Description: The percentage of time in hypoglycemia with blood glucose levels less than 54 mg/dL.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
percentage of time | 0.6 (2.2) | 0.2 (0.8)

8. Secondary Outcome: Percent of Time in Hyperglycemia (BG > 180 mg/dL)
Description: The percentage of time in hyperglycemia with blood glucose levels greater than 180 mg/dL.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
percentage of time | 49.1 (28.1) | 45.8 (30.7)

9. Secondary Outcome: Percent of Time in Hyperglycemia (BG>250 mg/dL)
Description: The percentage of time in hyperglycemia with blood glucose levels >250 mg/dL.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
percentage of time | 17.8 (22.8) | 16.5 (19.3)

10. Secondary Outcome: Number of Events of Prolonged Hypoglycemia
Description: The number of events of prolonged hypoglycemia, defined as > 1 and 2 hours, as determined by CGM.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: prologed hypoglycemia events
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
prologed hypoglycemia events
  Blood glucose <70 mg/dL | 0.12 (0.52) | 0.04 (0.29)
  Blood glucose <54 mg/dL | 0.12 (0.52) | 0.04 (0.29)

11. Secondary Outcome: Number of Hypoglycemia Events During the Day and Night
Description: The number of hypoglycemia events during the day and night in the POC testing group and the CGM-GTS group.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
events
  Blood glucose <70 mg/dL | 1.04 (2.72) | 1.70 (3.21)
  Blood glucose <54 mg/dL | 0.58 (2.00) | 0.64 (1.89)

12. Secondary Outcome: Number of Events of Hyperglycemia > 180 mg/dL
Description: Number of events of hyperglycemia > 180 mg/dL during the day and night between POC testing group and CGM-GTS group
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Count of Units; unit: blood glucose tests
Units Other Than Participants: blood glucose tests
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
Number analyzed (blood glucose tests) | 96 | 97
blood glucose tests | 77 | 96

13. Secondary Outcome: Number of Events of Hyperglycemia > 240 mg/dL
Description: Number of events of hyperglycemia > 240 mg/dL during the day and night between POC testing group and CGM-GTS group
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Count of Units; unit: blood glucose tests
Units Other Than Participants: blood glucose tests
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
Number analyzed (blood glucose tests) | 96 | 97
blood glucose tests | 54 | 75

14. Secondary Outcome: Percentage of POC BG Readings Within Target BG of 70 and 180 mg/dL
Description: The percentage of POC blood glucose readings within the target BG range of 70 and 180 mg/dL.
Time Frame: During hospitalization (up to 60 days of admission)
Population: POC data is unavailable for one participant in the POC study arm.
Measure: Mean (Standard Deviation); unit: percentage of tests
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 49 | 47
percentage of tests | 68 (33) | 61 (27)

15. Secondary Outcome: Glycemic Variability Calculated by Mean Amplitude of Glycemic Excursions (MAGE)
Description: Mean amplitude of glycemic excursions (MAGE), together with mean and standard deviation (SD), is the parameter for assessing glycemic variability and is calculated based on the arithmetic mean of differences between consecutive peaks and nadirs of differences greater than one SD of mean glycemia. It is designated to assess major glucose swings and exclude minor ones.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
mg/dL | 62.17 (24.0) | 64.03 (27.5)

16. Secondary Outcome: Number of Participants With Problems With Sensor Insertion
Description: The number of participants who experienced problems or issues while the sensor was being inserted was documented.
Time Frame: During hospitalization (up to 60 days of admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
Number analyzed (Participants) | 50 | 47
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time individuals gave consent to participate in the study and continued up to hospital discharge or for 60 days of admission (whichever came first).
Arm/Group | Point-of-care (POC) Testing With Blinded CGM (Standard of Care Study Arm) | Dexcom Continuous Glucose Monitoring (CGM) With Glucose Telemetry System (CGM-GTS)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/47
Other Adverse Events (participants affected / at risk) | 0/50 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT04818242/Prot_SAP_000.pdf